CLINICAL TRIAL: NCT03705338
Title: Elaboration of a Predictive Model in EEG for Induction and Emergence in Pediatric Patients Under General Anesthesia With Propofol
Brief Title: Predictive Model in EEG for Induction and Emergence in Pediatric With Propofol
Acronym: EEGPED
Status: Terminated | Type: Observational
Why Stopped: Outbreak COVID 19
Sponsor: Victor Contreras, MSN (Other)
Collaborators: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor-Investigator, Victor Contreras, MSN, Co-Investigator. Project Manager of Department of Anesthesiology, Pontificia Universidad Catolica de Chile
Organization: Pontificia Universidad Catolica de Chile (Other)
Other Study IDs: 180629004
Record Dates: First submitted 2018-10-05; First posted 2018-10-15 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-03

CONDITIONS: Electroencephalography; Anesthesia; Children, Only
Keywords: Anesthesia; Children; Electroencephalography; Propofol
MeSH Terms: interventions — Electroencephalography; Propofol; Anesthetics, General

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Electroencephalography: Electroencephalography (EEG) for induction and emergence in pediatric patients under general anesthesia with propofol.
  Interventions: Device: Electroencephalography; Drug: Propofol

INTERVENTIONS:
Device: Electroencephalography — Measure the appearance and disappearance of frontal alpha wave with EE, when them loss and recovery of consciousness under general anesthesia with propofol.
Drug: Propofol — Recorder the loss and recovery of consciousness in children under general anesthesia with TCI of propofol intravenous. Induction will be started with 20 mg/kg/hr of propofol up to UMSS level 4. Then will be titrated leading anesthesiologist criteria.
  Other Names: General anesthetic

SUMMARY:
Anesthesia is essential to control pain and produce unconsciousness during surgery and other procedures during childhood. The anesthetic deepness is measured indirectly through changes in blood pressure and heart rate or can be inferred according to estimated or measured concentrations of anesthetics.

In adults, anesthetic dosing, using patterns based on electroencephalogram (EEG) analysis, has shown clinical advantages compared to traditional monitoring. These advantages include lower consumption of hypnotics, less post-operative cognitive deterioration and decreased intraoperative awakening.

The maturation of the brain and Central Nervous System (CNS) that occurs in childhood affects the response of anesthetics. Additionally, the EEG changes with age and its dominant frequency is lower in children. This explains why brain monitoring methods developed in adults do not work well in children. However, these patterns cannot be extrapolated to the pediatric population. Therefore, it is necessary to develop indexes based on EEG with pediatric data to improve the dosage of hypnotics in this population.

The appearance of alpha wave in frontal EEG has been successfully used as a marker of unconsciousness during general anesthesia with GABAergic hypnotics in adults (sevoflurane, propofol). However, in children, the alpha wave appears since 4 months of age in anesthetics with sevoflurane, so studying the characterization of this wave during the loss and recovery of secondary consciousness anesthetic agents such as propofol has not been studied yet.

DETAILED DESCRIPTION:
Research question:

Is it possible to use the alpha wave as an indicator of loss and recovery of consciousness in anesthesia with propofol in children?

Hypothesis:

The appearance and disappearance of frontal alpha wave is a good indicator of loss and recovery of consciousness in anesthesia with propofol in children.

ELIGIBILITY:
Inclusion Criteria:

* ASA I - II
* Indications of phimosis surgery, cryptorchid and/or inguinal hernia surgery

Exclusion Criteria:

* Anatomical limitations for installing the EEG cap.
* Congenital or genetic malformations that influence his/her brain development.
* Neurological or cardiovascular disease
* Use of drugs with effect in the CNS in the last 24 hrs.
* Preterm newborn less than 32 weeks.

Ages: 3 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children with indications of surgery under general anesthesia and regional analgesia.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2021-10-15 (Actual)

PRIMARY OUTCOMES:
Loss and Recovery of consciousness | Continuously from start of propofol infusion to unarousable up to ending of infusion arouses without stimuli. In average 2 hrs.
  Recorded by the EEG signal - 40 channels waves: Beta, Alpha,Theta
Recovery of consciousness | From to ending of propofol infusion to arouses without stimuli. Continuously for 10 min.
  Watching the awakening and/or gross movement. Recorded by Go Pro cam the moment of Recovery of consciousness.
Loss of consciousness | From start of propofol infusion to unarousable to stimuli. Continuously for 10 min.
  Level 4 of University of Michigan Sedation Scale for children [0 0=awake/alert; 1=sleepy/responds appropriately; 2=somnolent/arouses to light stimuli ; 3=deep sleep/arouses to deeper physical stimuli; 4=unarousable to stimuli]. Recorded by Go Pro cam the moment of loss consciousness.

SECONDARY OUTCOMES:
Arterial Pressure | Entering operating room every 1 min per 5 min and every 5 min up to end of anesthesia or recovery of consciousness. In average 2 hrs.
  By non invasive Arterial Pressure: Systolic Arterial Pressure in mmHg, diastolic Arterial Pressure in mmHg and Medium Arterial Pressure in mmHg
Heart Rate | Entering operating room every 1 min per 5 min and every 5 min up to end of anesthesia or recovery of consciousness. In average 2 hrs.
  By EKG D-II bit per minute
Saturation Oxigen | Entering operating room every 1 min per 5 min and every 5 min up to end of anesthesia or recovery of consciousness. In average 2 hrs.
  Pulse Oximetry by reusable sensor in % of saturation.

CONTACTS AND LOCATIONS:
Overall Officials: Win Tin Chang, Principal Investigator — Pontificia Universidad Catolica de Chile
Locations (1):
- Victor Contreras, Santiago, Santiago Metropolitan, Chile

REFERENCES:
- [Background] Malviya S, Voepel-Lewis T, Tait AR, Merkel S, Tremper K, Naughton N. Depth of sedation in children undergoing computed tomography: validity and reliability of the University of Michigan Sedation Scale (UMSS). Br J Anaesth. 2002 Feb;88(2):241-5. doi: 10.1093/bja/88.2.241. PMID 11878656
- [Background] Cornelissen L, Donado C, Lee JM, Liang NE, Mills I, Tou A, Bilge A, Berde CB. Clinical signs and electroencephalographic patterns of emergence from sevoflurane anaesthesia in children: An observational study. Eur J Anaesthesiol. 2018 Jan;35(1):49-59. doi: 10.1097/EJA.0000000000000739. PMID 29120939
- [Background] Purdon PL, Pierce ET, Mukamel EA, Prerau MJ, Walsh JL, Wong KF, Salazar-Gomez AF, Harrell PG, Sampson AL, Cimenser A, Ching S, Kopell NJ, Tavares-Stoeckel C, Habeeb K, Merhar R, Brown EN. Electroencephalogram signatures of loss and recovery of consciousness from propofol. Proc Natl Acad Sci U S A. 2013 Mar 19;110(12):E1142-51. doi: 10.1073/pnas.1221180110. Epub 2013 Mar 4. PMID 23487781
- [Background] Brown EN, Purdon PL, Van Dort CJ. General anesthesia and altered states of arousal: a systems neuroscience analysis. Annu Rev Neurosci. 2011;34:601-28. doi: 10.1146/annurev-neuro-060909-153200. PMID 21513454
- [Background] Cornelissen L, Bergin AM, Lobo K, Donado C, Soul JS, Berde CB. Electroencephalographic discontinuity during sevoflurane anesthesia in infants and children. Paediatr Anaesth. 2017 Mar;27(3):251-262. doi: 10.1111/pan.13061. Epub 2017 Feb 8. PMID 28177176
- [Background] Cornelissen L, Kim SE, Purdon PL, Brown EN, Berde CB. Age-dependent electroencephalogram (EEG) patterns during sevoflurane general anesthesia in infants. Elife. 2015 Jun 23;4:e06513. doi: 10.7554/eLife.06513. PMID 26102526
- [Background] Fritz BA, Kalarickal PL, Maybrier HR, Muench MR, Dearth D, Chen Y, Escallier KE, Ben Abdallah A, Lin N, Avidan MS. Intraoperative Electroencephalogram Suppression Predicts Postoperative Delirium. Anesth Analg. 2016 Jan;122(1):234-42. doi: 10.1213/ANE.0000000000000989. PMID 26418126